CLINICAL TRIAL: NCT06719830
Title: Discrimination of Right Versus Left Septal Accessory Pathway Before and During the Electrophysiological Study
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwan Sayed Mahmoud, Lecturer of Cardiovascular Medicine, Assiut University
Other Study IDs: EPS for accessory pathway
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-09

CONDITIONS: WPW Syndrome; Accessory Pathway
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome; Pre-Excitation Syndromes | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Right group: Septal accessory pathway more to right
  Interventions: Procedure: Radiofrequency ablation
- Left group: Septal accessory pathway more to left
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — Radiofrequency ablation of the septal accessory pathway

SUMMARY:
Study of ECG and electrophysiological criteria which discriminate right versus left septal AP (both posteroseptal and anteroseptal AP). Both manifest and concealed APs will be considered .

DETAILED DESCRIPTION:
Radiofrequency catheter ablation is now the preferred treatment for patients with symptomatic Wolff-Parkinson-White (WPW) syndrome or recurrent symptomatic orthodromic reciprocating tachycardia . Successful ablation depends on the accurate localization of the accessory pathway (AP). Posteroseptal (inferior paraseptal) APs represent the second most common atrioventricular (AV) connection site after left free wall AP and often pose a diagnostic challenge. This is due to complex anatomy at the crux of the four cardiac chambers, where a small area may encompass APs that may be approached from the right or left endocardium, or require an epicardial ablation inside the coronary sinus (CS).

APs located in the posteroseptal area can take a variety of courses. Four different course types may be distinguished.

1. Endocardially between the inferior paraseptal right atrium and the right ventricle. This area includes the inferior part of the Koch's triangle and the area surrounding the CS ostium.
2. Endocardially between the inferior paraseptal left atrium and the left ventricle.
3. Coursing between the inferior paraseptal right atrium and the left ventricle in the pyramidal space, given that the right atrium lies directly on the posterior superior process of the left ventricle. This anatomical conformation results from the fact that the interatrial septum lies leftward to the interventricular septum and the tricuspid annulus is displaced 5-10 mm apically with respect to the mitral annulus. The right atrial endocardial aspect overlying the posterior superior process of the left ventricle lies between the most posterior aspect of the right fibrous trigone and the CS ostium, medial to the tricuspid valve. Because of its close proximity, ablation of these APs may be possible from the proximal CS.
4. Epicardially, connecting the musculature overlying the CS to the ventricle. These connections are related to sleeve-like extensions of the CS musculature that cover the proximal portion of the middle cardiac vein or posterior coronary veins. Most of these APs are ablated with a coronary venous These APs are referred to as 'epicardial CS' APs.

The procedural risks of inferior paraseptal AP ablation differ depending on whether a left-sided approach or a CS ablation is required .

Anteroseptal Aps are rare but associated with lower success rates and higher incidence of atrioventricular(AV) block. Anteroseptal AP can be ablated from right side , however Some including true para-Hisian APs can be safely and effectively ablated from the aortic cusps. Compared with the ablation at the right anteroseptal area, RF delivered at the aortic cusps has a higher immediate success, lower complication rate, and good long-term outcome. The aortic cusps should always be considered as the initial target for ablation of para-Hisian Aps . Data regarding the electro- cardiographic and electrophysiological characteristics as well as the safety and efficacy of catheter ablation of anteroseptal APs through the aortic cusps are limited Considering these differences, an accurate anticipation of location of septal AP is critical to inform the discussion and consent process with the patient and to guide the mapping strategy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with suggested septal AP (both manifest and concealed AP) undergoing electrophysiological study and ablation in EP cath lab in cardiology department, Assiut University Heart hospital.

Exclusion Criteria:

* Patients with redo AP or failed ablation.
* Patients with more than one AP.
* Congenital or structural heart diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with suggested septal AP (both manifest and concealed AP)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Differentiate right from left septal manifest accessory pathway using ECG | Baseline
  Onset of delta wave in each lead will be measured from the onset of the earliest delta wave in any of the ECG leads.The polarity of the delta wave will be measured within the initial 20 msec of the preexcitation and will be classified as positive (+), negative (-), or isoelectric (+-). Localization of the site of the accessory pathway will be done using Arruda's algorithm and Fitzpatrick's algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lebloa M, Pascale P. Preprocedural Discrimination of Posteroseptal Accessory Pathways Ablated from the Right Endocardium from Those Requiring a Left-sided or Epicardial Coronary Venous Approach. Arrhythm Electrophysiol Rev. 2022 Apr;11:e07. doi: 10.15420/aer.2021.55. PMID 35734142
- [Background] Jazayeri MR, Dhala A, Deshpande S, Blanck Z, Sra J, Akhtar M. Posteroseptal accessory pathways: an overview of anatomical characteristics, electrocardiographic patterns, electrophysiological features, and ablative therapy. J Interv Cardiol. 1995 Feb;8(1):89-101. doi: 10.1111/j.1540-8183.1995.tb00519.x. PMID 10155221
- [Background] Sealy WC, Mikat EM. Anatomical problems with identification and interruption of posterior septal Kent bundles. Ann Thorac Surg. 1983 Nov;36(5):584-95. doi: 10.1016/s0003-4975(10)60690-x. PMID 6639196
- [Background] Guiraudon GM, Klein GJ, Sharma AD, Jones DL, McLellan DG. Surgical ablation of posterior septal accessory pathways in the Wolff-Parkinson-White syndrome by a closed heart technique. J Thorac Cardiovasc Surg. 1986 Sep;92(3 Pt 1):406-13. PMID 3528678
- [Background] Sun Y, Arruda M, Otomo K, Beckman K, Nakagawa H, Calame J, Po S, Spector P, Lustgarten D, Herring L, Lazzara R, Jackman W. Coronary sinus-ventricular accessory connections producing posteroseptal and left posterior accessory pathways: incidence and electrophysiological identification. Circulation. 2002 Sep 10;106(11):1362-7. doi: 10.1161/01.cir.0000028464.12047.a6. PMID 12221053
- [Background] Calkins H, Yong P, Miller JM, Olshansky B, Carlson M, Saul JP, Huang SK, Liem LB, Klein LS, Moser SA, Bloch DA, Gillette P, Prystowsky E. Catheter ablation of accessory pathways, atrioventricular nodal reentrant tachycardia, and the atrioventricular junction: final results of a prospective, multicenter clinical trial. The Atakr Multicenter Investigators Group. Circulation. 1999 Jan 19;99(2):262-70. doi: 10.1161/01.cir.99.2.262. PMID 9892593
- [Background] Tai CT, Chen SA, Chiang CE, Lee SH, Chang MS. Electrocardiographic and electrophysiologic characteristics of anteroseptal, midseptal, and para-Hisian accessory pathways. Implication for radiofrequency catheter ablation. Chest. 1996 Mar;109(3):730-40. doi: 10.1378/chest.109.3.730. PMID 8617084
- [Background] Letsas KP, Efremidis M, Vlachos K, Georgopoulos S, Karamichalakis N, Saplaouras A, Xydonas S, Valkanas K, Sideris A. Catheter ablation of anteroseptal accessory pathways from the aortic cusps: A case series and a review of the literature. J Arrhythm. 2016 Dec;32(6):443-448. doi: 10.1016/j.joa.2016.02.010. Epub 2016 Apr 19. PMID 27920827
- [Background] Xu G, Liu T, Liu E, Ye L, Shehata M, Wang X, Li G. Radiofrequency catheter ablation at the non-coronary cusp for the treatment of para-hisian accessory pathways. Europace. 2015 Jun;17(6):962-8. doi: 10.1093/europace/euu271. Epub 2014 Oct 29. PMID 25355782
- [Background] Arruda MS, McClelland JH, Wang X, Beckman KJ, Widman LE, Gonzalez MD, Nakagawa H, Lazzara R, Jackman WM. Development and validation of an ECG algorithm for identifying accessory pathway ablation site in Wolff-Parkinson-White syndrome. J Cardiovasc Electrophysiol. 1998 Jan;9(1):2-12. doi: 10.1111/j.1540-8167.1998.tb00861.x. PMID 9475572
- [Background] Pambrun T, El Bouazzaoui R, Combes N, Combes S, Sousa P, Le Bloa M, Massoullie G, Cheniti G, Martin R, Pillois X, Duchateau J, Sacher F, Hocini M, Jais P, Derval N, Bortone A, Boveda S, Denis A, Haissaguerre M, Albenque JP. Maximal Pre-Excitation Based Algorithm for Localization of Manifest Accessory Pathways in Adults. JACC Clin Electrophysiol. 2018 Aug;4(8):1052-1061. doi: 10.1016/j.jacep.2018.03.018. Epub 2018 May 30. PMID 30139487
- [Background] Fitzpatrick AP, Gonzales RP, Lesh MD, Modin GW, Lee RJ, Scheinman MM. New algorithm for the localization of accessory atrioventricular connections using a baseline electrocardiogram. J Am Coll Cardiol. 1994 Jan;23(1):107-16. doi: 10.1016/0735-1097(94)90508-8. PMID 8277067